CLINICAL TRIAL: NCT04637932
Title: Use of Pro-seal LMA and Bronchoscopy During Percutaneous Dilatation Tracheostomy
Brief Title: Percutaneous Dilatation Tracheostomy, Broncoscopy, Pro-seal Laryngeal Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eylem Yaşar (Other)
Responsible Party: Sponsor-Investigator, Eylem Yaşar, Muğla Sıtkı Koçman Universty, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2020/60
Record Dates: First submitted 2020-11-03; First posted 2020-11-20 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Tracheostomy Complication
Keywords: percutan tracheostomy; bronchoscopy; pro-seal Laryngeal mask
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: Group 1 was determined as endotracheal tube and group 2 as pro-seal laryngeal mask group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of endotracheal tube During Percutaneous Dilatation Tracheostomy (Active Comparator): Group 1 was determined as endotracheal tube
  Interventions: Procedure: Percutaneous Dilatation Tracheostomy
- Use of Pro-seal LMA and Bronchoscopy During Percutaneous Dilatation Tracheostomy (Active Comparator): group 2 as pro-seal laryngeal mask group.
  Interventions: Procedure: Percutaneous Dilatation Tracheostomy

INTERVENTIONS:
Procedure: Percutaneous Dilatation Tracheostomy — pro-seal laryngeal mask or intubation tube in bronchoscopy-guided percutaneous dilation tracheostomy procedure.
  Other Names: Bronchoscopy

SUMMARY:
In this study, our primary goal is to compare whether there is any difference in the complication of using pro-seal laryngeal mask or intubation tube in bronchoscopy-guided percutaneous dilation tracheostomy procedure. Our secondary goal is to compare in terms of processing time.

DETAILED DESCRIPTION:
Following the approval of Muğla Sıtkı Koçman University Clinical Research Ethics Committee, 61 cases over the age of 18 who were scheduled for elective percutaneous dilatation tracheostomy in intensive care units were included in the study.

Elective percutaneous dilatation tracheostomy cases were randomly divided into two groups. Group 1 was determined as endotracheal tube and group 2 as pro-seal laryngeal mask group.

In the endotracheal tube group, which is a conventional method, after entering the trachea with percutaneous technique, the intubation tube was removed before dilatation and percutaneous dilatation tracheostomy was performed with the Seldinger method.

In the pro-seal laryngeal mask group, the fiberoptic bronchoscope was advanced with a pro-seal laryngeal mask, and after the correct position was achieved, percutaneous dilatation tracheostomy was performed using the Seldinger Method.

Arterial blood pressure, oxygen saturation, heart rate, arterial blood gas, mechanical ventilation mode, positive end expiratory pressure and mean airway pressure values were recorded before and 30 minutes after the procedure.

The time until the end of the procedure and complications were determined.

ELIGIBILITY:
Inclusion Criteria:hospitalized in intensive care units of our hospital and planned for elective percutaneous dilatation tracheostomy were included in the study.

-

Exclusion Criteria:

* history of cervical trauma,
* high-pressure mechanical ventilation (inspiratory pressure above 40 cmH2O),
* pulmonary edema,
* acute respiratory distress

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
complication of percutan dilatation tracheostomy procedure. | 7 days
  blood gas analysis, physical examination, lung auscultation, hemodynamics parameters

SECONDARY OUTCOMES:
processing time. | minutes
  Our secondary goal is to compare in terms of processing time.

CONTACTS AND LOCATIONS:
Overall Officials: semra Demirbilek, Study Director — Mugla Sitki Kocman University Department of AnesthesiaDepartment of Anesthesia
Locations (1):
- Mugla Sitki Kocman University, Muğla, Turkey (Türkiye)